CLINICAL TRIAL: NCT00515268
Title: A Double Blind, Placebo Controlled, Repeat Dose Study to Compare the Effectiveness of Two Doses of GSK256066 With Placebo in Reducing Lung Inflammation Following Segmental LPS Challenge in Healthy Volunteers
Brief Title: Endotoxin Challenge Study For Healthy Men and Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Diagnostic
Other Study IDs: IPC103711
Record Dates: First submitted 2007-08-09; First posted 2007-08-13 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: LPS challenge,; Healthy volunteers
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — 6-((3-((dimethylamino)carbonyl)phenyl)sulfonyl)-8-methyl-4-((3-methyloxyphenyl)amino)-3-quinolinecarboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subjects receiving GSK256066 (Experimental): Eligible subjects will be randomized to receive GSK256066 with inhaled doses of 25 micrograms or 87.5 micrograms once daily for 7 days, administered via an ACCUHALER.
  Interventions: Drug: GSK256066
- Subjects receiving placebo (Placebo Comparator): Eligible subjects will be randomized to receive placebo for 7 days, administered via an ACCUHALER.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK256066 — GSK256066 will be available as dry powder inhaler with dosing strengths of 12.5, 37.5, 50 micrograms per inhalation.
  Arms: Subjects receiving GSK256066
Drug: Placebo — Subjects will receive placebo inhaler.
  Arms: Subjects receiving placebo

SUMMARY:
The proposed study will examine the effect of pre-treatment with inhaled GSK256066 using a lung inflammation model induced by bronchoscopic instillation of bacterial endotoxin (lipopolysaccharide, LPS) in healthy volunteers.Data from this study will be used to support GSK256066 dose selection for future studies in COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females (contraception restrictions),
* 18-50yrs,
* BMI 19-31kg/m2,
* Non-smokers,
* FEV1 >/= 80% predicted

Exclusion Criteria:

* Abnormal troponin and/or CK MB,
* Participated in any GSK study involving the administration of COA for >/= 21 days.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2007-09-27 (Actual); Primary Completion 2008-04-23 (Actual); Study Completion 2008-04-23 (Actual)

PRIMARY OUTCOMES:
Absolute BAL neutrophils at 24 h post LPS exposure The total and differential cell count (absolute and percentage cell counts) in BAL at 24 h post LPS exposure | 24 hours

SECONDARY OUTCOMES:
Vital signs, ECG, FEV1, Serum concentration of protein inflammatory biomarkers, BAL concentrations of protein inflammatory biomarkers BAL concentrations of GSK256066, Day 1,Day 7&DAY 8 | Day 1,Day 7&DAY 8

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Hanover, Lower Saxony, Germany

REFERENCES:
- See also: Results for study IPC103711 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/IPC103711?search=study&study_ids=IPC103711#rs